CLINICAL TRIAL: NCT05012865
Title: Retrospective, Multicenter, Observational Study to Evaluate Current Treatment Outcomes in Japanese Patients With Metastatic Renal Cell Carcinoma Treated With Avelumab Plus Axitinib as a First-line Therapy
Brief Title: Current Treatment Outcomes in Japanese RCC Patients Treated With Avelumab Plus Axitinib as First-line Therapy: Retrospective Study (J-DART)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991043
Record Dates: First submitted 2021-07-26; First posted 2021-08-19 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Retrospective; Multicenter; Non-interventional; Medical chart review; Japan; Metastatic renal cell cancer(mRCC); Avelumab; Axitinib; First-line therapy; Standard care in real-world clinical setting
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — avelumab; Axitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with metastatic renal cell carcinoma: Patients with metastatic renal cell carcinoma
  Interventions: Drug: avelumab; Drug: axitinib

INTERVENTIONS:
Drug: avelumab — as provided in real world practice
Drug: axitinib — as provided in real world practice

SUMMARY:
This study is a multicenter, non-interventional, retrospective, medical chart review of patients with metastatic renal cell cancer(mRCC) treated with avelumab plus axitinib as a first-line therapy in Japan between 20 December 2019 and 20 December 2020. All decisions regarding clinical management and treatment of the participating patients were made by the investigator as part of standard care in real-world clinical setting and were not contingent upon the patient's participation in the study. Data will be collected if available per study site.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with metastatic renal cell cancer(mRCC) based on the General Rule for Clinical and Pathological Studies on Renal Cell Carcinoma (4th Edition) before receiving avelumab plus axitinib as a first-line therapy.
2. Over 20 years of age at the time of metastatic renal cell cancer(mRCC) diagnosis.
3. Start treatment with avelumab plus axitinib as a first-line therapy for metastatic renal cell cancer(mRCC) from 20 December 2019 to 20 December 2020.
4. For patients who are still alive and have routine visits to the study site, evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study. For patients who are still alive and had been transferred to another hospital, evidence that the patient has been informed of all pertinent aspects of the study and oral or written informed consent is obtained.
5. Deceased patients are also included for inclusion criteria 1-3.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic renal cell cancer(mRCC) treated with avelumab plus axitinib as a first-line therapy in Japan between 20 December 2019 and 20 December 2020
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - Kurume University Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Iwamizawa Municipal General Hospital, Iwamizawa, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - University Hospital,Kyoto Prefectural University of Medicine, Kamigyō-ku, Kyoto
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Jichi Medical University Saitama Medical Center, Saitama, Saitama
  - Hiroshima University Hospital, Hiroshima
  - Osaka City University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from participants with metastatic renal cell carcinoma (mRCC) who initiated treatment with avelumab plus axitinib as a first-line therapy in Japan, between 20-Dec-2019 and 20- Dec-2020 were included in this study. Data was retrieved and analyzed during approximately 4.5 months of this observational retrospective study.
Pre-assignment Details: All decisions regarding clinical management and treatment of the participants were made by the investigator as part of standard care in real-world clinical setting and were not dependent upon the participants' participation in the study.
Groups:
- Avelumab + Axitinib as First-line Therapy: Participants with mRCC treated with avelumab plus axitinib as a first-line therapy between 20-Dec-2019 to 20-Dec-2020 in Japan in real world practice. Participants were followed up to 20-Jun-2021 from index date (date of first prescription for avelumab plus axitinib between 20-Dec-2019 and 20 December 2020).
Period: Overall Study
Arm/Group | Avelumab + Axitinib as First-line Therapy
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included the medical records extracted for the purpose of the study from all eligible participants who were included in the study.
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized According to Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: ECOG-PS assessed participant's performance status on a 5 point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2= ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair. Participants whose score was not known were reported against "Unknown'.
Time Frame: Baseline (before first dose of avelumab plus axitinib, during data identification period from 20-Dec-2019 to 20-Dec-2020 [approximately 1 year]) retrieved data was analyzed during 4.5 months of this observational study
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  0 | 29
  1 | 9
  2 | 3
  3 | 0
  4 | 0
  Unknown | 7

2. Primary Outcome: Number of Participants Categorized According to International Metastatic RCC Database Consortium (IMDC) Risk Score
Description: IMDC criteria had 6 risk factors: Karnofsky Performance Status less than (<) 80% (ability to perform ordinary tasks, 0 [dead] -100 [normal]); time from diagnosis to start of systemic therapy <1 year; corrected serum calcium; neutrophils and platelets more than (>) upper limit of normal (ULN); hemoglobin <lower limit of normal (LLN). Present risk factors were added, and then participants were stratified as: favorable (0 factor), intermediate (1-2 factors), poor (more than or equal to [>=]3 factors).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Favorable | 8
  Intermediate | 26
  Poor | 14

3. Primary Outcome: Number of Participants Categorized According to Fuhrman Grade
Description: The four-tiered Fuhrman grading evaluates nuclear size, nuclear shape and presence of nucleolar prominence. Grade 1: small (=10 micrometer [mcm]) nuclear diameter, round/uniform nuclear shape and absent/inconspicuous nucleoli; Grade 2: large (=15 mcm) nuclear diameter, irregular outline nuclear shape and visible at *400 magnification nucleoli; Grade 3: larger (=20 mcm) nuclear diameter, obvious irregular outline nuclear shape and visible and prominent at *100 magnification nucleoli; Grade 4: grade 3 plus bizarre multilobed nuclei +/- spindle cells. Participants whose Fuhrman Grade were not known were reported against "Unknown'.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Grade 1 | 2
  Grade 2 | 14
  Grade 3 | 12
  Grade 4 | 8
  Unknown | 12

4. Primary Outcome: Number of Participants Categorized According to Histological Type
Description: In this outcome measure participants were reported according to the different histological type of mRCC including clear renal cell carcinoma, papillary renal cell carcinoma, chromophobe renal cell carcinoma and others.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Clear renal cell carcinoma | 39
  Papillary renal cell carcinoma | 1
  Chromophobe renal cell carcinoma | 1
  Others | 7

5. Primary Outcome: Number of Participants Categorized According to Presence of Sarcomatoid Component
Description: In this outcome measure, participants were categorized as "Yes" or "No" according to presence of sarcomatoid component were reported.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 5
  No | 43

6. Primary Outcome: Number of Participants Categorized According to Tumor-node-metastases (TNM) Classification
Description: TNM system is based on size of primary tumor (T), amount of spread to lymph nodes (N) and presence of metastases (M). T1: tumor <=20 millimeters (mm), T2: tumor >20 mm to <=50 mm, T3: >50 mm and TX: tumor cannot be assessed. N0: no lymph node metastases, N1: metastases to ipsilateral level I, II axillary lymph nodes, NX: Regional lymph nodes cannot be assessed. M0: no clinical/radiographic evidence of distant metastases, M1: distant detectable metastases as determined by clinical and radiographic means and/or histologically proven >0.2 mm, and MX: metastases cannot be assessed.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  T0 | 3
  T1 | 17
  T2 | 3
  T3 | 20
  T4 | 2
  TX | 3
  NX | 3
  N0 | 33
  N1 | 12
  MX | 2
  M0 | 6
  M1 | 40

7. Primary Outcome: Number of Participants Categorized According to Number of Metastatic Organs
Description: In this outcome measure participants were reported according to number of metastatic organs as a) 1 and, b) 2 or more.
Time Frame: as for outcome 1
Population: Full analysis set included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 43
Participants
  Metastatic organ 1 | 22
  Metastatic organs 2 or more | 21

8. Primary Outcome: Number of Participants Categorized According to Type of Site of Metastases
Description: Sites of metastases included: metastases of lung, liver, bone, brain, regional lymph nodes, distant nodal metastases and others. One participant could have more than 1 type of metastases.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 43
Participants
  Lung metastases | 25
  Liver metastases | 5
  Bone metastases | 14
  Brain metastases | 1
  Regional lymph node metastasis | 11
  Distant nodal metastasis | 4

9. Primary Outcome: Number of Participants According to Presence of Complications
Description: In this outcome measure participants were reported as "Yes" or "No" according to presence of complications.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 34
  No | 14

10. Primary Outcome: Number of Participants Who Underwent Nephrectomy Previously
Description: In this outcome measure, participants who underwent nephrectomy previously, were reported as "Yes' or "No".
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 32
  No | 16

11. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: GFR is an index of kidney function that describes the flow of filtered fluid through the kidney. eGFR was reported in millimeter per minute per 1.73 square meter (ml/min/1.73 m^2).
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 44
ml/min/1.73 m^2 | 49.62 (23.37)

12. Primary Outcome: Number of Participants With Proteinuria
Description: Proteinuria is the presence of an excess of serum proteins in the urine, which may be an early sign of kidney disease. Here, negative = <15 milligrams per deciliter (mg/dL), positive=15-29 mg/dL, 1 = 30 mg/dL, 2= 100 mg/dL, 3= 300 mg/dL.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 34
Participants
  Negative | 19
  Positive | 8
  1 | 3
  2 | 2
  3 | 2

13. Primary Outcome: C-reactive Protein (CRP)
Description: CRP was a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra-sensitive assay.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 44
Milligrams per deciliter | 1.779 (3.511)

14. Primary Outcome: Number of Participants Categorized According to Smoking Status
Description: In this outcome measure, participants with smoking history were reported as No (No smoking history, never smoked), No (Smoking history exists, quit smoking), Yes (currently smoking). Participant whose smoking status was not known were reported against "Unknown".
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  No (No smoking history) | 16
  No (Smoking history exists) | 21
  Yes | 5
  Unknown | 6

15. Primary Outcome: Number of Participants Who Took Concomitant Drugs
Description: In this outcome measure, participants who took concomitant drugs were reported.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 37
  No | 11

16. Secondary Outcome: Time to Treatment Failure (TTF) of Avelumab Plus Axitinib as a First-line Therapy
Description: TTF was defined as the time from the date of first dose of avelumab plus axitinib as first line therapy to the end of treatment for any cause earlier, including death. Kaplan-Meier method was used for analysis.
Time Frame: From index date up to 20-June-2021, where index date was date of first prescription for avelumab plus axitinib between 20-Dec-2019 and 20 December 2020 (maximum observation period was of 1.5 years approximately).
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Months | 15.2 [7.4 to NA] — Since participants with events were less hence upper limit of 95% CI could not be estimated.

17. Secondary Outcome: Real-world Progression Free Survival (PFS)
Description: PFS was defined as time from start of avelumab/axitinib treatment to date of first disease progression (DP) (as clinically assessed by local investigator based on radiology, laboratory evidence, pathology, or other assessments) or death due to any cause, whichever came first. If there were no clinical records of death or disease progression, they were censored at the date of initiation of the next line of therapy for the participants undertaking 2 or more lines of therapy based on the record, or at their last visit date during the study period for the participants undertaking only 1 line of therapy based on the record.
Time Frame: From avelumab plus axitinib initiation to disease progression or death due to any cause/censored date (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approx 1.6 years]); retrieved data was analyzed during 4.5 months of this OS
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Months | 15.3 [9.7 to NA] — Since participants with events were less hence upper limit of 95% CI could not be estimated.

18. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as percentage of participants with complete response (CR) or partial response (PR) as the best adjudication result in a method complied with RECIST version. 1.1 tumor assessment as closely as possible in clinical practice by investigator's judgment. CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30 percent (%) decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From avelumab plus axitinib initiation to CR or PR (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approximately 1.6 years]) retrieved data was analyzed during 4.5 months of this observational study
Population: Full analysis set included the medical records extracted for the purpose of the study from all eligible participants who were included in the study. "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and this time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 43
Percentage of participants | 48.8 [33.3 to 64.5]

19. Secondary Outcome: Time to Treatment Failure in Participants With Avelumab and Axitinib Treatment
Description: TTF was defined as the time from the date of first dose of avelumab plus axitinib to the end of treatment for any cause earlier, including death. Kaplan-Meier method was used for analysis.
Time Frame: From avelumab plus axitinib initiation to end of treatment (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approximately 1.6 years]) retrieved data was analyzed during 4.5 months of this observational study
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Months
  TTF: Avelumab | NA [5.4 to NA] — Since participants with events were less hence median and upper limit of 95% CI could not be estimated.
  TTF: Axitinib | 10.5 [3.9 to NA] — Since participants with events were less hence upper limit of 95% CI could not be estimated.

20. Secondary Outcome: Number of Participants With Discontinuation and Interruption of Avelumab and Axitinib Treatment
Description: In this outcome measure, number of participants who discontinued and had interruption of avelumab and axitinib treatment were reported.
Time Frame: From avelumab plus axitinib initiation to end of treatment (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approximately 1.6 years]); retrieved data was analyzed during 4.5 months of this observational study
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Avelumab: Discontinued | 8
  Avelumab: Interruption | 25
  Axitinib: Discontinued | 11
  Axitinib: Interruption | 28

21. Secondary Outcome: Number of Participants With Reason for Discontinuation of Avelumab Treatment
Description: In this outcome measure, participant who discontinued the avelumab treatment due to reasons including disease progression, adverse event, sufficient efficacy and others were reported. One participant could have more than 1 reason for discontinuation of treatment.
Time Frame: From avelumab plus axitinib initiation to end of treatment (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approximately 1.5 years]); retrieved data was analyzed during 4.5 months of this observational study
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 8
Participants
  Disease progression | 4
  Adverse event | 1
  Sufficient efficacy | 1
  Others | 3

22. Secondary Outcome: Number of Participants With Reason for Discontinuation of Axitinib Treatment
Description: In this outcome measure, participant who discontinued the axitinib treatment due to reasons including disease progression, adverse event, sufficient efficacy and others were reported. One participant could have more than 1 reason for discontinuation of treatment.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 11
Participants
  Disease progression | 3
  Adverse event | 3
  Sufficient efficacy | 2
  Others | 3

23. Secondary Outcome: Number of Participants With Reason for Interruption of Avelumab Treatment
Description: In this outcome measure, participant who had treatment interruption due to reasons including adverse event, sufficient efficacy and others were reported. One participant could have more than 1 reason for interruption of treatment.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 25
Participants
  Adverse event | 19
  Sufficient efficacy | 2
  Others | 10

24. Secondary Outcome: Number of Participants With Reason for Interruption of Axitinib Treatment
Description: as for outcome 23
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 28
Participants
  Adverse event | 24
  Sufficient efficacy | 2
  Others | 9

25. Secondary Outcome: Number of Participants With Dose Modification of Axitinib Treatment
Description: In this outcome measure, participants who had dose modification (increase/decrease) were reported.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 24
  No | 24

26. Secondary Outcome: Number of Participants According to Reason for Dose Modification of Axitinib Treatment
Description: In this outcome measure, number of participants were reported against the reasons for dose modification of axitinib treatment. One participant could have more than 1 reason for modification of axitinib treatment.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 24
Participants
  Adverse event | 19
  Others | 8

27. Secondary Outcome: Cumulative Dose of Corticosteroid for Immune-related Adverse Events (irAE) During Avelumab Plus Axitinib Treatment
Description: Immune-related adverse events (irAEs) was defined as the serious side effect of immune checkpoint inhibitor therapy for participants with advanced cancer.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 5
Milligrams
  Prednisolone: number analyzed (Participants) | 2
  Prednisolone | 15.00 (10.8)
  Methylprednisolone sodium succinate: number analyzed (Participants) | 2
  Methylprednisolone sodium succinate | 234.38 (110.5)
  Hydrocortisone sodium succinate: number analyzed (Participants) | 1
  Hydrocortisone sodium succinate | 50.00

28. Secondary Outcome: Duration of Corticosteroid Treatment for irAE During Avelumab Plus Axitinib Treatment
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 5
Days
  Prednisolone: number analyzed (Participants) | 2
  Prednisolone | 25.0 [14 to 172]
  Methylprednisolone sodium succinate: number analyzed (Participants) | 2
  Methylprednisolone sodium succinate | 1.0 [1 to 1]
  Hydrocortisone sodium succinate: number analyzed (Participants) | 1
  Hydrocortisone sodium succinate | 1.0 [1 to 1]

29. Secondary Outcome: Number of Corticosteroid Doses for irAE During Avelumab Plus Axitinib Treatment
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Number; unit: Doses
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 5
Doses
  Prednisolone: number analyzed (Participants) | 2
  Prednisolone | 2
  Methylprednisolone sodium succinate: number analyzed (Participants) | 2
  Methylprednisolone sodium succinate | 2
  Hydrocortisone sodium succinate: number analyzed (Participants) | 2
  Hydrocortisone sodium succinate | 1

30. Secondary Outcome: Number of Participants With Presence of Pre-medication for Potential Infusion-related Reaction of Avelumab
Description: In this outcome measure, number of participants who were on pre-medication and presence of these medications were reason for potential infusion-related reaction of avelumab, were reported.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 48
Participants
  Yes | 45
  No | 3

31. Secondary Outcome: Number of Participants Categorized According to Type of Pre-medication for Infusion-related Reaction of Avelumab
Description: In this outcome measure, number of participants who were on pre-medication and presence of these medications were reason for potential infusion-related reaction of avelumab, were reported according to type of pre-medications. One participant could have taken more than 1 type of pre-medication.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 45
Participants
  Acetaminophen | 39
  Chlorpheniramine maleate | 22
  Diphenhydramine hydrochloride | 22
  Famotidine | 4
  Diclofenac sodium | 1
  Hydrocortisone sodium succinate | 1
  Methylprednisolone sodium succinate | 1

32. Secondary Outcome: Number of Participants Who Received Treatment for Infusion-related Reaction of Avelumab
Description: In this outcome measure, number of participants who received any treatment for infusion-related reaction of avelumab were reported.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 45
Participants | 8

33. Secondary Outcome: Number of Participants by Type of Received Subsequent Treatment After Avelumab Plus Axitinib
Description: In this outcome measure, number of participants who received subsequent treatment after avelumab plus axitinib therapy, were reported according to type of subsequent treatment including tyrosine kinase inhibitors (TKI), immuno-oncology (IO) drugs and others. Categories with at least 1 non-zero data are reported below.
Time Frame: From avelumab plus axitinib end of treatment to end of study observation (during data identification period from 20-Dec-2019 to 20-Jun-2021 [approximately 1.5 years]); retrieved data was analyzed during 4.5 months of this observational study
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib as First-line Therapy
Number analyzed (Participants) | 12
Participants
  TKI: Pazopanib | 1
  TKI: Cabozantinib | 7
  IO: Nivolumab | 3
  Others: Axitinib + Pembrolizumab | 1

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected during the study
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event could not be met, hence safety data were not collected and reported.
Arm/Group | Avelumab + Axitinib as First-line Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05012865/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05012865/SAP_001.pdf